CLINICAL TRIAL: NCT00548808
Title: Comparison of Insulin Lispro Low Mixture With Insulin Glargine When Initiating and Intensifying Insulin Therapy As Required in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Oral Antihyperglycemic Medication
Brief Title: A Study for Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11541; F3Z-CR-IOPH (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin lispro low mixture (Experimental): Insulin lispro low mixture (1, 2 or 3 daily injections)
  Interventions: Drug: Insulin lispro low mixture
- Insulin glargine (Active Comparator): Insulin glargine (alone or with 1, 2 or 3 daily injections of insulin lispro)
  Interventions: Drug: Insulin glargine; Drug: Insulin lispro

INTERVENTIONS:
Drug: Insulin lispro low mixture — Dose depending on patient's need; subcutaneous injection before meal; start with once-daily injection before evening meal for 48 weeks, may add second injection before breakfast at any time during the treatment period if required, and may further add third injection before lunch at any time in the remainder of the treatment period if required.
  Other Names: LY275585[P]
  Arms: Insulin lispro low mixture
Drug: Insulin glargine — Dose depending on patient's need; one daily subcutaneous injection before bedtime for 48 weeks
  Arms: Insulin glargine
Drug: Insulin lispro — Dose depending on patient's need; subcutaneous injection before meal; may start once-daily injection before meal (e.g. lunch if the highest blood glucose value is measured before dinner) on top of insulin glargine at any time of the treatment period if required, and may further add second or even third injection in the remainder of the treatment period if required.
  Other Names: LY275585
  Arms: Insulin glargine

SUMMARY:
The purpose of the study is to compare the insulin lispro low mixture (1, 2 or 3 daily injections) with insulin glargine (alone or with 1, 2 or 3 insulin lispro daily injections) on lowering the blood sugar level

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Receiving oral antihyperglycemic medications (including metformin) without insulin injection in the last 90 days
* Hemoglobin A1c (HbA1c) equal to or greater than 7.0% but less than 11.0%
* Willing to receive insulin injection while continuing to take the prestudy oral antihyperglycemic medications
* Able to perform self monitoring of blood glucose

Exclusion Criteria:

* Are taking any other glucose-lowering agents other than metformin, sulfonylurea or Thiazolidinedione (Pioglitazone)
* Have taken acarbose, miglitol, pramlintide, exenatide, repaglinide, or nateglinide in the past 6 weeks, or for a total of 30 days or more, in the last 24 weeks
* Have a body mass index greater than 35 kg/m2
* History or presence of kidney disease
* Have cardiac disease (Class III or IV)

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM- 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daw Park, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Ringwood, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belém
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Campinas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mississauga, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottetown, Prince Edward Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
- India (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aligarh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbatore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyunggi-Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul

REFERENCES:
- [Derived] Bowering K, Reed VA, Felicio JS, Landry J, Ji L, Oliveira J. A study comparing insulin lispro mix 25 with glargine plus lispro therapy in patients with Type 2 diabetes who have inadequate glycaemic control on oral anti-hyperglycaemic medication: results of the PARADIGM study. Diabet Med. 2012 Sep;29(9):e263-72. doi: 10.1111/j.1464-5491.2012.03722.x. PMID 22672081
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients randomized but did not receive study drug: 1 withdrew, 1 did not want to use insulin, 1 lost to follow-up. Full Analysis Set: randomized, received at least 1 dose of study drug. Per-Protocol Set: randomized; no entry criteria violations; completed >=32 weeks of study; no systemic glucocorticoid therapy >14 cumulative days during study.
Groups:
- Insulin Lispro LM: Insulin lispro low mixture (1, 2 or 3 daily injections)
Period: Overall Study
Arm/Group | Insulin Lispro LM | Insulin Glargine
Started | 214 | 212
Full Analysis Set | 211 | 212
Per-Protocol Set | 177 | 184
Completed | 172 | 186
Not Completed | 42 | 26
Not completed — Lost to Follow-up | 9 | 3
Not completed — Protocol Violation | 8 | 8
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Physician Decision | 6 | 3
Not completed — Adverse Event | 4 | 5
Not completed — Death | 2 | 0
Not completed — Entry Criteria Not Met | 2 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Sponsor Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro LM | Insulin Glargine | Total
Number analyzed (Participants) | 211 | 212 | 423
Age Continuous [Mean (Standard Deviation); unit: years] | 56.68 (8.52) | 56.29 (9.35) | 56.48 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 107 | 225
  Male | 93 | 105 | 198
Race/Ethnicity, Customized [Number; unit: participants]
  African | 8 | 16 | 24
  Caucasian | 69 | 61 | 130
  East Asian | 78 | 77 | 155
  Hispanic | 35 | 36 | 71
  Native American | 1 | 0 | 1
  West Asian | 20 | 22 | 42
  West Asian (Indian sub-continent) | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 17 | 17 | 34
  Brazil | 33 | 34 | 67
  Canada | 28 | 28 | 56
  China | 29 | 30 | 59
  India | 53 | 53 | 106
  Korea, Republic of | 16 | 14 | 30
  Mexico | 35 | 36 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 48 Week Endpoint in Hemoglobin A1c (HbA1c)
Time Frame: Baseline, 48 weeks
Population: Per-protocol set: randomized, no entry criteria violations, completed >=32 weeks of study, and no systemic glucocorticoid therapy for >14 cumulative days during study. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percent (%) glycated hemoglobin
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 177 | 184
percent (%) glycated hemoglobin | -1.91 (0.23) | -1.87 (0.23)
Statistical Analysis 1: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 0.4% for HbA1c was used; p = 0.716, ANCOVA; ANCOVA Model: Change in HbA1c = Treatment + Baseline + Country + Sulfonylurea use (Type III sums of squares); Least Squares Mean Difference = -0.04, 95% CI 2-sided [-0.25 to 0.17], Standard Error of Mean 0.11 — Least Squares Mean Difference = Insulin Lispro LM minus Insulin Glargine

2. Secondary Outcome: Change in Hemoglobin A1c (HbA1c) Over Time
Time Frame: Baseline, 16 Weeks, 32 Weeks, 48 Weeks
Population: Per-protocol set: randomized, no entry criteria violations, completed >=32 weeks of study, and no systemic glucocorticoid therapy for >14 cumulative days during study.
Measure: Least Squares Mean (Standard Error); unit: percent (%) glycated hemoglobin
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 177 | 184
percent (%) glycated hemoglobin
  16 Week Change from Baseline | -1.65 (0.23) | -1.76 (0.23)
  32 Week Change from Baseline | -1.92 (0.23) | -1.90 (0.23)
  48 Week Change from Baseline | -1.91 (0.23) | -1.87 (0.23)
Statistical Analysis 1: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.279, Mixed Models Analysis — P-value for 16 Week Change from Baseline; Mixed Model Analysis: Change in HbA1c = Treatment + Baseline + Country + Sulfonylurea use + Visit + Treatment*Visit (Type 3 sums of squares)
Statistical Analysis 2: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.846, Mixed Models Analysis — P-value for 32 Week Change from Baseline; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.741, Mixed Models Analysis — P-value for 48 Week Change from Baseline; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Patients Achieving HbA1c <6.5% and <7% Over Time
Time Frame: 16 weeks, 32 weeks, 48 weeks
Population: Per-protocol set: randomized; no entry criteria violations; completed >=32 weeks of study; no systemic glucocorticoid therapy >14 cumulative days during study.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 177 | 184
percentage of participants
  Percent achieving HbA1c < 6.5 % at 16 weeks | 10.2 | 12.5
  Percent achieving HbA1c < 7.0 % at 16 weeks | 28.2 | 32.6
  Percent achieving HbA1c < 6.5 % at 32 weeks | 19.4 | 17.5
  Percent achieving HbA1c < 7.0 % at 32 weeks | 40.6 | 38.8
  Percent achieving HbA1c < 6.5 % at 48 weeks | 21.2 | 19.0
  Percent achieving HbA1c < 7.0 % at 48 weeks | 40.0 | 39.1
Statistical Analysis 1: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.465, Regression, Logistic — P-value for patients achieving HbA1c <6.5% at 16 weeks; Generalized Estimating Equation model with fixed effects for treatment, country, sulfonylurea use, baseline HbA1c, visit, and visit*treatment; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.41 to 1.50]
Statistical Analysis 2: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.365, Regression, Logistic — P-value for Patients Achieving HbA1c <7% at 16 Weeks; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.51 to 1.28]
Statistical Analysis 3: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.683, Regression, Logistic — P-value for patients achieving HbA1c <6.5% at 32 weeks; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.65 to 1.95]
Statistical Analysis 4: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.810, Regression, Logistic — P-value for patients achieving HbA1c <7% at 32 weeks; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.68 to 1.64]
Statistical Analysis 5: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.555, Regression, Logistic — P-value for patients achieving HbA1c <6.5% at 48 weeks; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.69 to 2.01]
Statistical Analysis 6: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.829, Regression, Logistic — P-value for patients achieving HbA1c <7% at 48 weeks; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.67 to 1.64]

4. Secondary Outcome: 7-point Self-monitored Blood Glucose Profiles
Time Frame: Baseline, 16 weeks, 32 weeks, 48 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 177 | 184
millimoles per liter (mmol/L)
  Morning Pre-Meal Baseline | 9.92 (2.28) | 10.04 (2.36)
  Morning Postprandial Meal Baseline | 13.64 (3.13) | 13.70 (3.42)
  Midday Pre-Meal Baseline | 10.36 (3.22) | 10.62 (3.12)
  Midday Postprandial Meal Baseline | 12.77 (2.91) | 12.70 (3.36)
  Evening Pre-Meal Baseline | 10.39 (2.72) | 10.65 (3.14)
  Evening Postprandial Meal Baseline | 12.59 (3.09) | 12.80 (3.64)
  0300 Hours Baseline | 10.09 (2.82) | 10.12 (3.03)
  Morning Pre-Meal Week 16 | 7.04 (1.84) | 6.55 (1.67)
  Morning Postprandial Meal Week 16 | 9.79 (2.74) | 9.55 (2.79)
  Midday Pre-Meal Week 16 | 7.94 (2.37) | 7.64 (2.33)
  Midday Postprandial Meal Week 16 | 10.13 (2.63) | 9.58 (2.65)
  Evening Pre-Meal Week 16 | 8.52 (2.50) | 7.81 (2.46)
  Evening Postprandial Meal Week 16 | 9.35 (2.73) | 9.80 (2.90)
  0300 Hours Week 16 | 7.15 (2.09) | 7.01 (1.96)
  Morning Pre-Meal Week 32 | 6.62 (1.55) | 6.21 (1.19)
  Morning Postprandial Meal Week 32 | 8.80 (2.43) | 8.73 (2.09)
  Midday Pre-Meal Week 32 | 6.93 (2.12) | 6.90 (1.76)
  Midday Postprandial Meal Week 32 | 9.33 (2.49) | 8.86 (2.14)
  Evening Pre-Meal Week 32 | 7.71 (2.18) | 7.50 (1.92)
  Evening Postprandial Meal Week 32 | 8.62 (2.26) | 8.96 (2.31)
  0300 Hours Week 32 | 6.63 (1.75) | 6.75 (1.73)
  Morning Pre-Meal Week 48 | 6.74 (1.52) | 6.37 (1.17)
  Morning Postprandial Meal Week 48 | 8.79 (2.28) | 8.85 (2.21)
  Midday Pre-Meal Week 48 | 7.01 (1.99) | 6.99 (1.79)
  Midday Postprandial Meal Week 48 | 9.25 (2.31) | 8.88 (2.31)
  Evening Pre-Meal Week 48 | 7.33 (1.86) | 7.33 (2.03)
  Evening Postprandial Meal Week 48 | 8.74 (2.11) | 8.90 (2.29)
  0300 Hours Week 48 | 6.53 (1.54) | 6.56 (1.73)

5. Secondary Outcome: Change From Baseline in Postprandial Blood Glucose Over Time
Description: The change in blood glucose was evaluated by the GlycoMark™ test. GlycoMark measures levels of 1,5 anhydroglucitol (1,5 AG) in serum or plasma, allowing for the short- to intermediate-term monitoring of glycemic control in patients with diabetes. When 1,5 AG values decrease, serum glucose levels increase.
Time Frame: Baseline, 16 weeks, 32 weeks, 48 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 177 | 184
millimoles per liter
  Week 16 Change from Baseline | 3.32 (1.16) | 3.55 (1.17)
  Week 32 Change from Baseline | 4.69 (1.19) | 4.56 (1.18)
  Week 48 Change from Baseline | 5.24 (1.20) | 4.89 (1.20)
Statistical Analysis 1: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.604, Mixed Models Analysis — P-value for Week 16 Change from Baseline; Mixed Model Analysis: Change in Blood Glucose = Treatment + Baseline + Country + HbA1c stratum + Sulfonylurea use + Visit + Treatment*Visit
Statistical Analysis 2: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.814, Mixed Models Analysis — P-value for Week 32 Change from Baseline; [statistical method as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.582, Mixed Models Analysis — P-value for 48 Week Change from Baseline; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Daily Total Insulin Dose (U/Day) at 16, 32, and 48 Weeks
Time Frame: 16 weeks, 32 weeks, 48 weeks
Population: Full Analysis Set: all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units of insulin per day (U/day)
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 211 | 212
Units of insulin per day (U/day)
  Week 16 | 36.42 (25.90) | 35.87 (21.55)
  Week 32 | 50.38 (34.02) | 48.16 (31.18)
  Week 48 | 54.97 (37.12) | 54.03 (35.90)

7. Secondary Outcome: Daily Total Insulin Dose Per Body Weight (U/kg/Day) at 16, 32, and 48 Weeks
Time Frame: 16 weeks, 32 weeks, 48 weeks
Population: Full Analysis Set: all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units of insulin/kilogram/day (U/kg/day)
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 211 | 212
Units of insulin/kilogram/day (U/kg/day)
  Week 16 | 0.49 (0.36) | 0.49 (0.29)
  Week 32 | 0.65 (0.43) | 0.65 (0.42)
  Week 48 | 0.71 (0.45) | 0.71 (0.47)

8. Secondary Outcome: Change From Baseline to 48 Week Endpoint in Lipid and Cholesterol Profiles
Time Frame: baseline, 48 weeks
Population: Full Analysis Set: all randomized participants who received at least one dose of study drug and had baseline and endpoint values.
Measure: Least Squares Mean (Standard Error); unit: millimoles/Liter (mmol/L)
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 211 | 212
millimoles/Liter (mmol/L)
  Cholesterol (n=195, n=203) | -0.18 (0.18) | -0.08 (0.18)
  Triglycerides (n=195, n=203) | -0.09 (0.21) | 0.03 (0.21)
  Low Density Lipoprotein (n=178, n=191) | -0.11 (0.17) | -0.06 (0.17)
  High Density Lipoprotein (n=195, n=203) | 0.06 (0.05) | 0.04 (0.05)
Statistical Analysis 1: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.162, ANCOVA — P-value for Cholesterol; ANCOVA model: Lab Result = Treatment + Baseline + Country + HbA1c stratum + Sulfonylurea use (Type III sums of squares); Least Squares Mean Difference = -0.11, 95% CI 2-sided [-0.26 to 0.04], Standard Error of Mean 0.08 — Least Squares Mean Difference = Insulin Lispro LM minus Insulin Glargine
Statistical Analysis 2: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.165, ANCOVA — P-value for Triglycerides; ANCOVA model: Lab Result = Treatment + Baseline + Country + HbA1c stratum + Sulfonylurea use (Type III sums of squares); Least Squares Mean Difference = -0.12, 95% CI 2-sided [-0.30 to 0.05], Standard Error of Mean 0.09 — Least Squares Mean Difference = Insulin Lispro LM minus Insulin Glargine
Statistical Analysis 3: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.510, ANCOVA — P-value for Low Density Lipoprotein; ANCOVA model: Lab Result = Treatment + Baseline + Country + HbA1c stratum + Sulfonylurea use (Type III sums of squares); Least Squares Mean Difference = -0.05, 95% CI 2-sided [-0.18 to 0.09], Standard Error of Mean 0.07 — Least Squares Mean Difference = Insulin Lispro LM minus Insulin Glargine
Statistical Analysis 4: Comparison: Insulin Lispro LM vs Insulin Glargine; Test type: Superiority or Other; p = 0.382, ANCOVA — P-value for High Density Lipoprotein; ANCOVA model: Lab Result = Treatment + Baseline + Country + HbA1c stratum + Sulfonylurea use (Type III sums of squares); Least Squares Mean Difference = 0.02, 95% CI 2-sided [-0.02 to 0.06], Standard Error of Mean 0.02 — Least Squares Mean Difference = Insulin Lispro LM minus Insulin Glargine

9. Secondary Outcome: Safety: Number of Participants With Serious and Non-Serious Adverse Events
Description: Safety was assessed via serious adverse events (SAEs) and AEs, the details of which are listed in the Reported Adverse Event section.
Time Frame: baseline through 48 weeks
Population: Full Analysis Set: all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro LM | Insulin Glargine
Number analyzed (Participants) | 211 | 212
participants
  Serious Adverse Events | 19 | 13
  Non-Serious Adverse Events | 107 | 116

ADVERSE EVENTS:
Arm/Group | Insulin Lispro LM | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 19/211 | 13/212
Other Adverse Events (participants affected / at risk) | 107/211 | 116/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro LM (N=211) | Insulin Glargine (N=212)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) — One of these events resulted in death.
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0) — This event resulted in death.
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro LM (N=211) | Insulin Glargine (N=212)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Cataract (Eye disorders) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 5 (7)
Gastritis (Gastrointestinal disorders) | 4 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 10 (11) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 8 (8)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Furuncle (Infections and infestations) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 17 (24) | 22 (28)
Localised infection (Infections and infestations) | 1 (1) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 4 (5)
Nasopharyngitis (Infections and infestations) | 13 (15) | 9 (11)
Pharyngitis (Infections and infestations) | 4 (5) | 2 (2)
Respiratory tract infection (Infections and infestations) | 3 (4) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 7 (9)
Urinary tract infection (Infections and infestations) | 10 (11) | 10 (10)
Viral infection (Infections and infestations) | 0 (0) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 8 (8) | 4 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (8)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 4 (4)
Headache (Nervous system disorders) | 8 (14) | 3 (4)
Sciatica (Nervous system disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Hypertension (Vascular disorders) | 8 (8) | 9 (9)
Venous insufficiency (Vascular disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days